CLINICAL TRIAL: NCT04670783
Title: Measuring the Efficacy of Surgical and Percutaneous Neuroablative Procedures in the Management of Plateaued or Refractory Upper-extremity Spasticity.
Brief Title: Surgery and Neuroablative Procedures in Spasticity
Status: Completed | Type: Observational
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Mahdis Hashemi, Research Assistant, Vancouver Island Health Authority
Other Study IDs: H2019-03232
Record Dates: First submitted 2020-11-17; First posted 2020-12-17 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Upper Extermity Spasticity; Multidisciplinary Approach; Novel Algorithm; Diagnostic Nerve Block; Surgery; Percutaneous Neuroablative Procedures; Refractory Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — Orthopedic surgery (i.e. tenotomy, tendon transfer) or percutaneous neuroablative procedures (i.e. cryoneurotomy) which will be done for upper limb refractory spasticity after being triaged by DNB.
  Other Names: Percutaneous neuroablation

SUMMARY:
For many patients with spasticity, traditional therapies have not achieved maximal outcomes. Due to common complaints such as pain, limb positioning and hygiene concerns, there has been an increase demand for other adjunctive therapies like surgeries and other interventions. This spasticity multidisciplinary clinic consisting of a physiatrist, plastic surgeon and anesthesiologist is performing a novel approach to refractory spasticity to triage and designed a treatment plan for them as routine medical care. This study will document the efficacy of this novel designed multidisciplinary approaches for intervention in complex spasticity patients, and will develop a decision-making algorithm in spasticity including both traditional treatment (i.e. botulinum toxin , bracing) and novel treatments(i.e. neurectomy , cryoneurotomy).

DETAILED DESCRIPTION:
Many patients continue to live with disabling spasticity that negatively affects their health, independence and quality of life. For these patients, traditional therapies such as bracing, medications, and botulinum toxin have not achieved maximal outcomes. Up to one-quarter of physicians have noted to be limited by the maximal dosage of botulinum toxin allowed in their country. Due to common complaints of pain, difficulty with limb positioning, and hygiene concerns there has been an increase in demand for novel adjunctive therapies, including surgery, to improve patient outcomes.

The deisgned triage pathway is based on the diagnostic lidocaine nerve block (DNB), which is already using in Franco-European studies and has been accepted as academic abstract at the Canadian Association of Physical Medicine and Rehabilitation Annual Meeting in Gatineau Quebec in 2019. In this approach, patients are triaged for intervention based on their responses to DNB, which is applying local anesthesia to a selected nerve branch. Also the investigators of this study who have created Canada's first interdisciplinary spasticity clinic consisting of a physiatrist, plastic surgeon and anesthesiologist are working to bring the world-leading spasticity interventions to Canada and developing Canadian techniques. This includes cryoneurotomy and selective microfascicular neurectomy. Both of these techniques have been developed in this multidisciplinary clinic and in the past three years and have been published as journal articles, academic posters or presented at international congresses.This research is a pilot study to test the present current triage and treatment pathways. This study will evaluate the patients with upper limb spasticity who are going to have any of traditional treatments (i.e. bracing, botulinum toxin) or novel treatments (i.e. cryoneurotomy, tenotomy, neurotomy) as their standard medical cares. All these assessments are parts of their standard evaluations and the available data will be collected for this study. These data include their range of motions, spasticity grades, upper limb function, pain, satisfaction and injected botulinum toxin dosage. These data will be used to document the efficacy of this approach by comparing these measurements that are already done for their standard clinical care. Also, the final result will be helpful to create a Canadian algorithm to approach patients with refractory upper limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years old, with upper extremity spasticity causing functional impairment.
* Patients that have plateaued in outcomes in which the clinical examination suggests further interventions can be trialed.
* The clinical examination, including a V1 (maximal passive stretch) and V3 (Fast catch) on upper extremity examination that demonstrates further passive or active range may be possible, versus if contracture must be managed. For example, a fisted hand that can be forced open. This includes factors such as fluctuating tone or clonus interfering with the assessment.
* The patient undergoes a diagnostic nerve block to determine if there is reducible spasticity in the muscle versus contracture.
* The patient has been offered a neuroablative procedure or surgery and has elected to undergo the procedure. The patient has consented to undergo the said procedure.

Exclusion Criteria:

* Patients where no consent or Assent is obtained
* Unable to attend treatment schedule,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient with upper limb spasticity who has been triaged to have surgery or neuroablative procedure after undergoing a successful DNB.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Degree of changes in spasticity as assessed by Modified Ashworth Scale from baseline and in 1, 3, 6, 9 and 12 months after the intervention. | up to 12 months after intervention
  The test will be done by the trained assistant which is not enrolled in providing medical care. The scale has 5 grades and based on severity of spasticity the examiner will assign a number to each tested movement. The grades are shown as 0, 1, 1+, 2, 3, 4. In grade 0 patient shows no spasticity , while grade 4 means maximum spasticity and the affected limb is rigid in flexion or extention.
Degree of changes in range of motion of tested joints as assessed by Tardieu Scale from base line and in 1, 3, 6, 9 and 12 months. | up to 12 months
  The maximum of passive range of motion in slow movement(V1) and degree of catch in speed (V3) and active range of motion will be measured by goniometer.
Upper limb function changes as assessed by Disabilities of the Arm, Shoulder and Hand questionnaire ( DASH questionnaire)(2006). | up to 12 months
  It is a self-administered questionnaire that participants will be asked to fill out at baseline and in 1, 3, 6, 9 and 12 months. Final score will be calculated based on the provided formula and will be between (0) , which means patient has no difficulty at all and (100) which means the worst outcome.
Patients satisfaction in achieving their goals after the procedure as assessed by Patients satisfaction in achieving their goals after the procedure as assessed by Goal Attainment Scale. | up to 12 months after procedure
  Patients satisfaction in achieving their goals after the procedure as assessed by Goal Attainment Scale38. Based on this scale participants will be asked for 3 main goals that they desire to achieve after the intervention. The baseline score will be (-1) and they will be interviewed again at 1, 3, 6, 9 and 12 months, to record how they reported their achievement. The scores of (-2), (-0.5), (0), (+1) and (+2) will be assigned if they feel that their condition is worst than before, better but not as good as expected, as expected, better than expected and much better than expected. All goals will be weighted equally, and final score will be calculated based on the available formula, in each session. The higher score is presenting of better outcome

SECONDARY OUTCOMES:
Upper limb function changes as assessed by Box and Block test. | up to 12 months after procedure.
  Participants will be in sitting position and will be asked to move the cubes from one part to the other part in 1 minute.The test will be done in baseline and in 1, 3,6, 9 and 12 months.
Changes in pain as assessed by Brief Pain Inventory Questionnaire. | up to 12 months
  This is a self-administered questionnaire that will be provided for participants for filing out at baseline and in 1, 3, 6, 9 and 12 months after the intervention.The Patient will ask to answer each question by choosing a number between 0 to 10, and the final score is calculating by adding these numbers together and then divided by 4. The result will show the severity of patient pain out of 10. (0 means no pain and 10 means the worst pain that can be imagine)
Changes in hand resting position as assessed by Keenan Scale. (the name of the physician that first described that in 1987) | 12 months after intervention
  Changes in the Hand resting position as assessed by Keenan Scale. Participants will be assessed by an independent examiner and based on available scale their hand position will be graded. Grade 1 is the minimum deformity while grade 5 Is the maximum deformity which is presented by clenched fist and palmar hygiene problem. The assessment will be done at baseline and in 1, 3, 6, 9 and 12 months.
Changes in thumb position as assessed by House Scale (The name of physician that first described this classification in 1981). | 12 months after the procedure
  Changes in thumb deformity (position of thumb in relation to other fi ngers) as assessed by House Scale (1981).Participants will be assessed by an independent examiner and based on available scale their thumb position will be graded between 1 to 4. Grade 1 is the minimum deformity and 4 is the maximum deformity. The assessment will be done at baseline and in 1, 3, 6, 9 and 12 months.
Changes in hand function as assessed by House Functional Scale ( the name of the physician that first described this scale in 1981). | up to 12 months after intervention
  The test will be done by an independent examiner and participants will be asked to pick a cube on the table while they are in a sitting position. Based on the available scale (o= No movement and 8= spontaneous use, complete) their hand function will be graded in baseline, 1,3,6,9 and 12 months after intervention.
Changes in hand grip strength as assessed by dynamometer from baseline to 1,3,6,9 and 12 months. | up to 12 months after the intervention
  The test will be done by Jamar Dynamometer and will be recorded as kilogram.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Winston, MD FRCPC, Principal Investigator — VIHA
Locations (1):
- Victoria General Hospital, Victoria, British Colombia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wissel J, Verrier M, Simpson DM, Charles D, Guinto P, Papapetropoulos S, Sunnerhagen KS. Post-stroke spasticity: predictors of early development and considerations for therapeutic intervention. PM R. 2015 Jan;7(1):60-7. doi: 10.1016/j.pmrj.2014.08.946. Epub 2014 Aug 27. PMID 25171879
- [Background] Bensmail D, Hanschmann A, Wissel J. Satisfaction with botulinum toxin treatment in post-stroke spasticity: results from two cross-sectional surveys (patients and physicians). J Med Econ. 2014 Sep;17(9):618-25. doi: 10.3111/13696998.2014.925462. Epub 2014 Jun 12. PMID 24841450
- [Background] Yelnik AP, Hentzen C, Cuvillon P, Allart E, Bonan IV, Boyer FC, Coroian F, Genet F, Honore T, Jousse M, Fletcher D, Velly L, Laffont I; SOFMER group; SFAR group; Viel E. French clinical guidelines for peripheral motor nerve blocks in a PRM setting. Ann Phys Rehabil Med. 2019 Jul;62(4):252-264. doi: 10.1016/j.rehab.2019.06.001. Epub 2019 Jun 13. PMID 31202956
- [Background] Winston P, Mills PB, Reebye R, Vincent D. Cryoneurotomy as a Percutaneous Mini-invasive Therapy for the Treatment of the Spastic Limb: Case Presentation, Review of the Literature, and Proposed Approach for Use. Arch Rehabil Res Clin Transl. 2019 Oct 17;1(3-4):100030. doi: 10.1016/j.arrct.2019.100030. eCollection 2019 Dec. PMID 33543059
- [Background] Winston P, Krauss E, Vincent D. Cryoneurotomy of the bilateral lateral pectoral nerves in a quadriplegic patient with spasticity, a novel approach. ISPRM 2020 Poster. 2020.
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] House JH, Gwathmey FW, Fidler MO. A dynamic approach to the thumb-in palm deformity in cerebral palsy. J Bone Joint Surg Am. 1981 Feb;63(2):216-25. PMID 7462278
- [Derived] Winston P, MacRae F, Rajapakshe S, Morrissey I, Boissonnault E, Vincent D, Hashemi M. Analysis of Adverse Effects of Cryoneurolysis for the Treatment of Spasticity. Am J Phys Med Rehabil. 2023 Nov 1;102(11):1008-1013. doi: 10.1097/PHM.0000000000002267. Epub 2023 Apr 24. PMID 37104641

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04670783/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04670783/ICF_000.pdf